CLINICAL TRIAL: NCT01526902
Title: Proclear 1-D Multifocal Nondispensing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-12-02A
Record Dates: First submitted 2012-02-02; First posted 2012-02-06 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-03

CONDITIONS: Presbyopia
Keywords: contact lenses
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- omafilcon A / PC 1-D MF (Active Comparator): omafilcon A (PC 1-D MF) / lotrafilcon B (AIR OPTIX MF)
  Subjects were randomly assigned into either the omafilcon A/PC 1-D MF lenses with +0.75D over-correction in the non-dominant eye or the lotrafilcon B/Air Optix MF lenses then crossed-over into the alternative pair of study lenses.
  Interventions: Device: omafilcon A / PC 1-D MF; Device: lotrafilcon B / Air Optix MF
- lotrafilcon B / Air Optix MF (Active Comparator): lotrafilcon B (AIR OPTIX MF) / omafilcon A (PC 1-D MF)
  Subjects were randomly assigned into either the omafilcon A/PC 1-D MF lenses with +0.75D over-correction in the non-dominant eye or the lotrafilcon B/Air Optix MF lenses then crossed-over into the alternative pair of study lenses.
  Interventions: Device: omafilcon A / PC 1-D MF; Device: lotrafilcon B / Air Optix MF

INTERVENTIONS:
Device: omafilcon A / PC 1-D MF — Subjects were randomly assigned into either the omafilcon A/PC 1-D MF lenses with +0.75D over-correction in the non-dominant eye or the lotrafilcon B/Air Optix MF lenses then crossed-over into the alternative pair of study lenses.
  Other Names: Proclear Multifocal daily wear soft contact lenses
Device: lotrafilcon B / Air Optix MF — Subjects were randomly assigned into either the omafilcon A/PC 1-D MF lenses with +0.75D over-correction in the non-dominant eye or the lotrafilcon B/Air Optix MF lenses then crossed-over into the alternative pair of study lenses
  Other Names: Air OPtix Aqua Multifocal extended wear soft contact lenses

SUMMARY:
This study is designed to compare the relative performance related to subjective and objective vision between two multifocal soft contact lenses.

DETAILED DESCRIPTION:
The aim of this study was to compare the subjective and objective vision. of Proclear® 1-D Multifocal test lenses (MF) with +0.75D overcorrection of the distance lens power in the nondominant eye compared to the Air Optix® Aqua Multifocal (CIBA VISION) contact lenses in low, Medium and High Add presbyopic subjects (+1.25 to +2.50 inclusive).

ELIGIBILITY:
Inclusion Criteria:

* Be between 40 and 65 years of age (inclusive)
* Require a reading addition of +1.25 to +2.50D (inclusive)
* Spherical distance CL or spectacle prescription between +3.00D and -5.00D(inclusive)
* Spectacle cylinder less than or equal to 0.75D in both eyes.
* Currently has a reading add correction in their spectacle or CL habitual correction (e.g. if myope, removes distance correction to read)
* Normal binocularity (no amblyopia, no strabismus, no habitually uncorrected anisometropia ≥ 2.00D)
* Have a minimum 2 weeks soft contact lens experience
* Be able to wear the study lens (e.g. good fit is attained and acceptable subjective comfort and vision for the duration of the study)
* Able to read, comprehend and sign an informed consent
* Willing to comply with the wear and study visit schedule
* Monocular best-corrected distance visual acuity ≥ 20/25 in each eye
* No gas permeable contact lens wear for 1 month prior to the study

Exclusion Criteria:

To be eligible for the study, each candidate must not present with any of the following

* Any active corneal infection, injury, inflammation, or ocular abnormality
* Systemic or ocular allergies, which might interfere with contact lens wear
* Systemic disease, which might interfere with contact lens wear
* Ocular disease, which might interfere with contact lens wear
* Pregnant or lactating
* Strabismus/amblyopia
* Habitually uncorrected anisometropia greater than or equal to 2.00 D
* Subjects who have undergone corneal refractive surgery
* Subjects with keratoconus or other severe corneal irregularity contraindicating lens wear

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kollbaum, OD, PhD, Principal Investigator — Clinical Optics Research Lab, Indiana University, Bloomington, Indiana, USA
Locations (1):
- Clinical Optics Research Lab, Indiana University,, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was open between 06FEB2012 and 28FEB2012
Pre-assignment Details: The subjects who are current contact lens wearers should attend the first visit wearing their habitual lenses and having worn them that day for at least 2 hours prior to the visit.
Groups:
- Omafilcon A (PC 1-D MF) / Lotrafilcon B (AIR OPTIX MF); Lotrafilcon B (AIR OPTIX MF) / Omafilcon A (PC 1-D MF): Subjects were randomly assigned into either the omafilcon A (PC 1-D) Multifocal with +0.75D over-correction in the non-dominant eye or the Air Optix Aqua (lotrafilcon B)Multifocal lenses as their initial pair. Lens Pair 1 were evaluated for fit, vision and comfort (1 hour after lens application). Following this evaluation and during this same visit, the subject then crossed-over into the alternative pair of study lenses. This second pair of lenses was also evaluated for fit, vision and comfort (1 hour after lens application).
Period: Overall Study
Arm/Group | Omafilcon A (PC 1-D MF) / Lotrafilcon B (AIR OPTIX MF) | Lotrafilcon B (AIR OPTIX MF) / Omafilcon A (PC 1-D MF)
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: Subjects were randomly assigned into either the omafilcon A/PC 1-D MF lenses with +0.75D over-correction in the non-dominant eye or the lotrafilcon B/Air Optix MF lenses then crossed-over into the alternative pair of study lenses.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Objective Vision Assessments: High Contrast Distance Visual Acuity
Description: Tested with charts distant to the subject with both eyes together in normal lighting conditions. The unit of measure is logMAR units (logarithm of the minimum angle of resolution) A logMAR acuity of 0.0 equates to 20/20 Snellen acuity. Positive logMAR values indicate poorer vision and negative values denote better visual acuity than baseline 20/20 value.
Time Frame: After 1 hour of lens wear
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: logMAR units
Groups:
- PC1DMF: (Test Lens) omafilcon A Proclear 1-D multifocal lens
- Air Optix MF: (Control Lens) lotrafilcon B Air Optix Aqua Multifocal
Arm/Group | PC1DMF | Air Optix MF
Number analyzed (Participants) | 49 | 49
logMAR units | -0.09 (0.08) | -0.05 (0.08)

2. Secondary Outcome: Subjective Overall Vision: High Contrast Distance Visual Quality
Description: Subjects instructed to rate Vision quality at distance, intermediate and near vision (OU) using a 0-100 numerical scale where 0 = poor and 100 = excellent.
Time Frame: After 1 hour of lens wear
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PC1DMF | Air Optix MF
Number analyzed (Participants) | 49 | 49
units on a scale | 87 (16) | 88 (11)

3. Secondary Outcome: Subjective Vision Assessments: High Contrast Intermediate Visual Quality
Description: as for outcome 2
Time Frame: After 1 hour of lens wear
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PC1DMF | Air Optix MF
Number analyzed (Participants) | 49 | 49
units on a scale | 85 (15) | 85 (15)

4. Primary Outcome: Objective Vision Assessments: High Contrast Intermediate Visual Acuity
Description: Tested with charts at intermediate distance (100cm)distant to the subject with both eyes together in normal lighting conditions. The unit of measure is logMAR units (logarithm of the minimum angle of resolution) A logMAR acuity of 0.0 equates to 20/20 Snellen acuity. Positive logMAR values indicate poorer vision and negative values denote better visual acuity than baseline 20/20 value.
Time Frame: After 1 hour of lens wear
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: logMAR units
Arm/Group | PC1DMF | Air Optix MF
Number analyzed (Participants) | 49 | 49
logMAR units | -0.11 (0.08) | -0.10 (0.09)

5. Primary Outcome: Objective Vision Assessments: High Contrast Near Visual Acuity
Description: Tested with charts set at near point (40cm)distant to the subject with both eyes together in normal lighting conditions. The unit of measure is logMAR units (logarithm of the minimum angle of resolution) A logMAR acuity of 0.0 equates to 20/20 Snellen acuity. Positive logMAR values indicate poorer vision and negative values denote better visual acuity than baseline 20/20 value.
Time Frame: After 1 hour of lens wear
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: logMAR units
Arm/Group | PC1DMF | Air Optix MF
Number analyzed (Participants) | 49 | 49
logMAR units | 0.08 (0.14) | 0.05 (0.12)

6. Secondary Outcome: Subjective Vision Assessments: High Contrast Near Visual Quality
Description: as for outcome 2
Time Frame: After 1 hour of lens wear
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PC1DMF | Air Optix MF
Number analyzed (Participants) | 49 | 49
units on a scale | 81 (18) | 80 (18)

ADVERSE EVENTS:
Groups:
- Omafilcon A / PC1DMF L2A (TEST); Lotrafilcon B / Air Optix MF (CONTROL): Low-Med and High Add power groups were randomly assigned to either omafilcon A/Proclear Multifocal soft contact lenses (PC1DMF L2A) or lotrafilcon B/Air OPtix Aqua Multifocal soft contact lenses (Air Optix MF) then crossed-over into the alternative pair of study lenses.
Arm/Group | Omafilcon A / PC1DMF L2A (TEST) | Lotrafilcon B / Air Optix MF (CONTROL)
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days